CLINICAL TRIAL: NCT05397119
Title: A Ph1 Randomized Double-Blind Controlled Dose-Range Safety Tolerability & Immunogenicity Study of 2 Doses of Intranasal rH5 Flu Vaccine With & Without Nanoemulsion Adjuvant Followed by 1 Boost of Intramuscular H5N1 Vaccine in Healthy Adults
Brief Title: A Safety and Immunogenicity of Intranasal Nanoemulsion Adjuvanted Recombinant Pandemic Flu Vaccine in Healthy Adults
Acronym: IN-NE-rH5
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BlueWillow Biologics (Industry)
Collaborators: University of Maryland, Baltimore (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BW-1014-001; U01AI148081 (NIH); 20-0036 (Other: DMID Protocol Number)
Record Dates: First submitted 2022-05-13; First posted 2022-05-31 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Influenza, Pandemic
Keywords: Pandemic influenza; Nanoemulsion adjuvant; Nasal vaccine; rH5
MeSH Terms: conditions — Influenza, Human | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive BW-1014 in 3 different dose levels (25 µg, 50 µg or 100 µg rH5 in NE adjuvant), using a pipette dropper. Control arms include rH5 alone (without NE adjuvant) or placebo (saline) control.
  Since this is first in humans, a dose escalation assessment will take place. A sentinel group of 2 participants from the lowest dose (25 µg rH5 in NE) with 2 rH5 control and 2 placebo control will be dosed first before proceeding to the next dose level. Each escalation of dose will take place after safety clearance of the prior lower dose level. Dosing of the remainder of subjects per dose arm will take place after safety clearance of the corresponding dose sentinel participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All IN study vaccines are milky white in appearance. Vaccinators will be unblinded to vaccine allocation, but they will have no role in assessment of vaccine safety or immunogenicity. Only the vaccine compounding personnel, the unblinded vaccinator, and the study statistician will have access to the randomization code prior to study completion. Unblinding procedures are described in the Manual of Operations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BW-1014: 25 µg rH5 in 20% NE - pipette - IN (Experimental): 20% Nanoemulsion and 25 µg recombinant H5 antigen administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Interventions: Biological: BW-1014: 25 µg rH5 in 20% NE - pipette - IN; Biological: H5N1 IIV - IM
- BW-1014: 50 µg rH5 in 20% NE - pipette - IN (Experimental): 20% Nanoemulsion and 50 µg recombinant H5 antigen administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Interventions: Biological: BW-1014: 50 µg rH5 in 20% NE - pipette - IN; Biological: H5N1 IIV - IM
- BW-1014: 100 µg rH5 in 20% NE - pipette - IN (Experimental): 20% Nanoemulsion and 100 µg recombinant H5 antigen administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Interventions: Biological: BW-1014: 100 µg rH5 in 20% NE - pipette - IN; Biological: H5N1 IIV - IM
- rH5 (100 µg) control - pipette - IN (Placebo Comparator): 100 µg recombinant H5 antigen (without adjuvant) administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Interventions: Biological: rH5 (100 µg) control - pipette - IN; Biological: H5N1 IIV - IM
- Saline (Placebo) - pipette - IN (Sham Comparator): Saline (negative control) administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Interventions: Biological: Saline (Placebo) - pipette - IN; Biological: H5N1 IIV - IM

INTERVENTIONS:
Biological: BW-1014: 25 µg rH5 in 20% NE - pipette - IN — 20% Nanoemulsion and 25 µg recombinant H5 antigen administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Arms: BW-1014: 25 µg rH5 in 20% NE - pipette - IN
Biological: BW-1014: 50 µg rH5 in 20% NE - pipette - IN — 20% Nanoemulsion and 50 µg recombinant H5 antigen administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Arms: BW-1014: 50 µg rH5 in 20% NE - pipette - IN
Biological: BW-1014: 100 µg rH5 in 20% NE - pipette - IN — 20% Nanoemulsion and 100 µg recombinant H5 antigen administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Arms: BW-1014: 100 µg rH5 in 20% NE - pipette - IN
Biological: rH5 (100 µg) control - pipette - IN — 100 µg recombinant H5 antigen (without adjuvant) administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Arms: rH5 (100 µg) control - pipette - IN
Biological: Saline (Placebo) - pipette - IN — Saline (negative control) administered intranasally by an electronic pipette (500µL) Two doses administered 4 weeks apart
  Arms: Saline (Placebo) - pipette - IN
Biological: H5N1 IIV - IM — 90 µg H5N1 IIV administered intramuscularly (1 mL) One booster dose administered 6 months following last immunization

SUMMARY:
The purpose of this clinical trial is to evaluate the safety and immunogenicity of BW-1014.

BW-1014 is a nanoemulsion (NE) adjuvanted recombinant Hemagglutinin 5 (rH5) that would protect against pandemic flu.

The study will be conducted in 40 healthy adults volunteers, age 18 - 45, in one center in the United States.

The study will compare 3 different dose levels of rH5 (25µg, 50µg and 100µg rH5 in 20% NE adjuvant using a pipette dropper with rH5 control (100µg without NE adjuvant) and placebo control (saline). The investigational product will be administered in 2 doses intranasally (IN). This will be followed 6 months later with a licensed H5N1 IIV IM vaccine.

In addition to safety outcome, homologous and heterologous immunological outcomes will be tested in nasal wash, serum, and blood cells.

DETAILED DESCRIPTION:
This study is a single center, phase 1, first-in-human, single-center, randomized, placebo-controlled, double-blind study to assess the safety, tolerability, and immunogenicity of a primary series of intranasal recombinant H5 influenza vaccine with and without nanoemulsion adjuvant followed by boosting dose of licensed, intramuscular influenza A (H5N1) vaccine.

Participants will be randomized in one of the following 5 arms:

A. BW-1014: 25 µg / 20% NE; 8 participants. B. BW-1014: 50 µg / 20% NE; 8 participants. C. BW-1014: 100 µg / 20% NE; 8 participants. D. rH5 control: 100µg; 8 participants. E. Saline (Placebo); 8 participants. Because this is a dose escalation trial, our study has four stages with one cohort receiving vaccines at each stage. Up to 40 participants will be randomized to one of the five study groups at an allocation ratio depending on the escalation stage. If all participants proceed to vaccination, the final vaccine allocation ratio will be 1:1:1:1:1. Subjects will receive a primary series of two intranasal vaccinations of study treatment administered on Days 1 and 29. Subject dosing will proceed in a stepwise process. Each dose of adjuvanted study vaccine will be assessed in sentinel participants before the remainder of the study group is vaccinated and before proceeding to vaccination of sentinel participants with the next higher dose of adjuvanted study vaccine. Following receipt of the first vaccine dose, sentinel participants will be followed for 7 days for halting criteria and SMC data review prior to proceeding with vaccination of the remainder of the study group. All participants will subsequently receive a third dose of intramuscular, heterologous influenza A (H5N1) vaccine on Day 197.

Participants will be followed for safety and immunology endpoints for one year following their second study treatment vaccination.

Participants will be assessed for production of specific mucosal and humoral antibodies in addition to cellular immune response in mononuclear cells collected from peripheral blood and from nasal wash fluid throughout the study. These assessments will be to both homologous H5N1 clade 2.1 and heterologous H5N1 clade 1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women aged 18 through 45 years of age, inclusive.
2. Women must not be pregnant or nursing. If premenopausal, absence of pregnancy must be confirmed by a negative serum pregnancy test conducted at screening and a negative urine pregnancy test conducted at the site within 24 hours preceding receipt of vaccine.
3. Women who are not surgically sterile or at least one year post-menopausal must agree to use acceptable birth control. Acceptable birth control methods include oral, implantable, transdermal or injectable contraceptive; barrier methods such as condoms, cervical caps, or diaphragms with spermicide; abstinence from sexual relationships with a male partner, non-male sexual relationships, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the first study vaccination, and other reliable forms of contraception approved by the Investigator. Acceptable birth control must be used for a minimum of 30 days prior to vaccination and for 3 months following final study vaccination.
4. Subjects must be in good general health, as determined by medical history and physical examination. Acceptable vital signs and clinical laboratory examinations are within the normal range per study toxicity tables (Appendix B). Vital signs and clinical laboratory examinations meeting Grade 1 criteria may also be acceptable in the opinion of the PI or appropriate Sub-Investigator. For this study, an appropriate Sub-Investigator is a designated clinician licensed to make medical diagnoses and listed on the Form FDA 1572. Exclusionary clinical laboratory examinations may be repeated one time to assess clinical improvement in the event temporary halting criteria (described in Section 8.6.2) are met at the time of the first examination.
5. Subjects must be able to comprehend the study requirements as evidenced by a score of ≥ 70% on the comprehension assessment (two attempts permitted), be available for the required study period, and have the ability to attend scheduled visits.
6. Subjects must be able to provide written informed consent to participate in the study.
7. Subject agrees to future use of left-over specimens and to the collection of additional specimens for potential future use research.
8. Receipt of the CDC-recommended number of doses of an EUA authorized or licensed COVID-19 vaccine product ≥ four weeks prior to first study vaccination.

Exclusion Criteria:

1. Presence of significant acute or chronic, uncontrolled medical or psychiatric illness (institution of new medical or surgical treatment, or a significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months). This includes signs or symptoms consistent with upper or lower respiratory tract infections.
2. Participants with symptoms of COVID-19 and/or who are positive for SARS-CoV-2 by molecular testing conducted within 2 days prevaccination.
3. Have known hypersensitivity or allergy to eggs, egg or chicken protein, or other components of the Influenza Virus Vaccine, H5N1 (Sanofi Pasteur).
4. Receipt of licensed or experimental H5N1 influenza vaccine ever.
5. Subjects with a history of chronic cough, frequent sinus infections, sinusitis, allergic rhinitis, nasal polyps or obstruction, including deviated septum significant enough to obstruct the nasal openings or a history of nasal surgery.
6. Body mass index (BMI) BMI ≤ 18.5 or ≥ 40.
7. Positive serology for human immunodeficiency virus (HIV)-1 or HIV-2, hepatitis B, or hepatitis C (HCV).
8. Platelet count less than 100,000/mm prior to randomization during baseline visit.
9. History of drug or chemical abuse within the past year prior to screening.
10. History of aspiration, dysphagia, swallowing disorders, stroke or other neurologic conditions that may predispose the subject to aspiration of test articles into the respiratory tract.
11. History of Bell's palsy.
12. History of Guillain-Barré syndrome within 6 weeks of prior influenza virus vaccine.
13. Cancer or treatment for cancer, within 3 years. Basal cell carcinoma or squamous cell carcinoma are allowed, unless present on or near the nose.
14. Impaired immune responsiveness, including a history of diabetes mellitus.
15. Chronic use of inhaled or intranasal sprays including decongestants and corticosteroids.
16. A current vaper, smoker or tobacco user or a history of smoking or tobacco use within the past year prior to screening.
17. Receipt or history of receiving any medications or treatments that affected the immune system such as immune globulin, interferon, immunomodulators, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids (oral or injectable) in the past 6 months.
18. Has received or has plans to receive any licensed or authorized vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to first study vaccination through Day 57.
19. History of allergic and/or anaphylactic type reaction to injected influenza vaccines or to any of the components of BW-1014 [soybean oil, dehydrated alcohol (anhydrous ethanol), polysorbate (Tween 80), cetylpyridinium chloride (CPC), and tobacco].
20. Receipt of any investigational product or nonregistered drug within the 30 days before screening or currently enrolled in any investigational drug study or intends to enroll in such a study within the ensuing 13-month period.
21. Use of nasally administered prescription or over-the-counter medications within 7 days before vaccination.
22. Receipt of blood or blood products 8 weeks before screening or planned administration prior to the Week 8 visit.
23. Donation of blood or blood products within 8 weeks before screening or at any time up to the Week 4 clinic visit.

If a subject presents at screening or on a vaccination date with an acute illness, the Investigator will refer to Individual Halting Criteria to assess whether to temporarily delay enrollment or vaccination until the illness is resolved.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-10-12 (Actual); Study Completion 2023-10-12 (Actual)

PRIMARY OUTCOMES:
Safety Outcome: Number of participants reporting local or systemic reactions | Up to Day 29
  Local and systemic reactions will be assessed in the clinic within 1 hour of intranasal BW-1014, positive control, and placebo administration, including visual assessment of nasal passages
Safety Outcome: Number of participants reporting solicited reactions and general AEs | Up to Day 36
  Solicited reactions and general AEs will be assessed in follow up visit/phone call within 7 days of vaccination with intranasal BW-1014, positive control and placebo
Safety Objective: Number of participants reporting unsolicited AEs | Up to Day 57
  Unsolicited AEs will be assessed in follow up visits/phone calls within 28 days of primary vaccinations with intranasal BW-1014, positive control and placebo
Safety Outcome: Number of participants reporting any hematological and biochemical laboratory abnormality (Class 1 of higher) | Up to Day 43
  Hematological and biochemical laboratory abnormality (Class 1 of higher) will be assessed in follow up visits within 7 days of first dose intranasal BW-1014 or within 14 days second dose intranasal BW-1014, positive control, and placebo
Safety Outcome: Number of participants reporting medically attended AEs (MAAEs) | Up to Day 57
  MAAEs will be assessed in follow up visits/phone calls within 28 days of primary vaccinations with intranasal BW-1014, positive control, and placebo
Safety Outcome: Number of participants reporting serious adverse events (SAEs) | Up to Day 393
  SAEs will be assessed by study arm. An adverse event is considered "serious" if it results in death, or a life-threatening AE, or in hospitalization, or in a substantial disruption of the ability to conduct normal life functions, or in a congenital anomaly/birth defect.
Safety Outcome: Number of participants reporting potential immune-mediated medical conditions (PIMMCs) | Up to Day 393
  PIMMCs will be assessed by follow up visits/phone calls following vaccinations with intranasal BW-1014, positive control, and placebo
Safety Outcome: Number of participants reporting new onset chronic medical conditions (NOCMCs) | Up to Day 393
  NOCMCs will be assessed by follow up visits/phone calls following vaccinations with intranasal BW-1014, positive control, and placebo

SECONDARY OUTCOMES:
Safety endpoint: Number of participants reporting local or systemic reactions to intramuscular H5N1 IIV vaccine | Day 197
  Local or systemic reactions will be assessed within 1 hour of vaccination with intramuscular H5N1 IIV vaccine
Safety endpoint: Number of participants reporting solicited reactions and general AEs | Day 204
  Solicited reactions and general AEs will be assessed within 7 days of vaccination with intramuscular H5N1 IIV vaccine
Safety endpoint: Number of participants reporting unsolicited AEs | Day 225
  Unsolicited AEs will be assessed within 28 days of vaccinations with intramuscular H5N1 IIV vaccine
Safety endpoint: Number of participants reporting any hematological and biochemical laboratory abnormality (Class 1 of higher) | Day 204
  Hematological and biochemical laboratory abnormality (Class 1 of higher) will be assessed within 7 days of vaccination with intramuscular H5N1 IIV vaccine,
Safety endpoint: Number of participants reporting medically attended AEs (MAAEs) | Day 225
  MAAEs will be assessed within 28 days of vaccination with intramuscular H5N1 IIV vaccine,
Primary Humoral Immune Response Outcome: HI Geometrical Mean Titers levels | Up to Day 57
  The primary humoral immune response to homologous H5N1 (clade 2.1) will be measured using hemagglutinin inhibition assays after two doses of intranasal vaccine or placebo
Primary Humoral Immune Response Outcome: Rates of seroconversion | Day 57 compared to Day 1
  Rates of seroconversion are defined as the percentage of subjects with either a pre-vaccination HI titer < 1:10 and a post-vaccination HI titer > 1:40 or a pre-vaccination HI titer > 1:10 and a minimum of four-fold rise in post-vaccination HI antibody titer.
Primary Humoral Immune Response Outcome: IgA and IgG endpoint titer levels | Up to Day 57
  Strain-specific GMT by ELISA will be measured using ELISA after two doses of intranasal vaccine or placebo
Primary Mucosal Immunogenicity Outcome: Mucosal vaccine-specific IgA Geometric Mean Titer (GMT) | Up to Day 197
  Mucosal vaccine-specific IgA Geometric Mean Titer (GMT) will be assessed by ELISA
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific activation marker (CD69), cytokines/chemokines | Up to Day 197
  Vaccine-specific activation marker (CD69) will be assessed in cells isolated from the nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific activation marker (CD154), cytokines/chemokines | Up to Day 197
  Vaccine-specific activation marker (CD154) will be assessed in cells isolated from the nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal vaccine-specific IgG Geometric Mean Titer (GMT) | Up to Day 197
  Mucosal vaccine-specific IgG Geometric Mean Titer (GMT) will be assessed by ELISA
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific IFN-gamma | Up to Day 197
  Vaccine-specific cytokine (IFN-gamma) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific TNF-α | Up to Day 197
  Vaccine-specific cytokine (TNF-α) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific IL-4 | Up to Day 197
  Vaccine-specific cytokine (IL-4) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific IL-2 | Up to Day 197
  Vaccine-specific cytokine (IL-2) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific IL-10 | Up to Day 197
  Vaccine-specific cytokine (IL-10) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific IL-21 | Up to Day 197
  Vaccine-specific cytokine (IL-21) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific CD107a | Up to Day 197
  Vaccine-specific degranulation marker (CD107a) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific Granzyme B | Up to Day 197
  Vaccine-specific degranulation marker (Granzyme B) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific T-cell memory subset (effector memory cell) | Up to Day 197
  Vaccine-specific T-cell memory subset (effector memory cell) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific T-cell memory subset (central memory cell) | Up to Day 197
  Vaccine-specific T-cell memory subset (central memory cell) will be assessed in cells isolated from nasal cavity by Flow Cytometry
Primary Mucosal Immunogenicity Outcome: Mucosal Vaccine-specific T-cell memory subset (effector memory CD45RA+ cell) | Up to Day 197
  Vaccine-specific T-cell memory subset (effector memory CD45RA+ cell) will be assessed in cells isolated from nasal cavity by Flow Cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ortiz, MD, MS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Center for Vaccine Development and Global Health, University of Maryland School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deming ME, Toapanta FR, Pasetti M, Golding H, Khurana S, Hamouda T, Fattom A, Liang Y, Tennant SM, McGilvray MF, Bernal PJ, Oshinsky JJ, Datta S, Booth JP, Coughlan L, Neuzil KM, Costley CD, Kotloff KL, Sztein MB, Ortiz JR; rH5 Writing Group. An intranasal adjuvanted, recombinant influenza A/H5 vaccine primes against diverse H5N1 clades: a phase I trial. Nat Commun. 2025 Nov 6;16(1):9321. doi: 10.1038/s41467-025-64686-3. PMID 41198655